CLINICAL TRIAL: NCT03309865
Title: A Pilot Study Evaluating the Synergistic Effect of Vedolizumab in Conjunction With Structured Semi-Vegetarian Diet on the Treatment of Ulcerative Colitis.
Brief Title: Evaluating the Combined Effect of Vedolizumab and Semi-Vegetarian Diet on Ulcerative Colitis.
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Not enough patients to enroll.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ming-Hsi Wang, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 17-005613
Record Dates: First submitted 2017-10-07; First posted 2017-10-16 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Ulcerative Colitis; Dietary Modification
Keywords: semi-vegetarian diet; vedolizumab; ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined diet and vedolizumab (Experimental): Intervention: vedolizumab injection (300mg, IV infusions at week 0, 2, 6, 14) and concurrently on structured semi-vegetarian diet; Duration of Therapy: 14 weeks
  Interventions: Dietary Supplement: semi-vegetarian diet; Drug: Vedolizumab Injection

INTERVENTIONS:
Dietary Supplement: semi-vegetarian diet — semi-vegetarian dietary intervention: Duration of Therapy: 14 weeks;
Drug: Vedolizumab Injection — vedolizumab (300mg) IV infusions at week 0, 2, 6, 14; Duration of Therapy: 14 weeks
  Other Names: vedolizumab

SUMMARY:
Research of fecal microflora and dysbiosis status in ulcerative colitis (UC) has shown its influential role on the disease pathogenesis. Vedolizumab, a humanized monoclonal antibody blocking the migration of leukocytes into inflamed intestinal tissue, has been shown to achieve remission in about half of active UC patients. Dietary intervention in UC patients has not been adequately studied. There is a significant clinical gap to achieve a higher efficacy and better clinical outcomes on the treatment of active UC patients. This study proposes to assess the integrated effect of normalization of intestinal dysbiosis through a structured semi-vegetarian dietary intervention in active UC patients who will also be under the standard of care medical therapy (vedolizumab).

Significance of investigation for innovation: The pathogenesis of UC has been found to be multi-factorial, including host genetics and dysregulated inflammatory response, and recent research has shown the influential role of gut environmental factors - dysbiosis which has been found the key feature of UC. Vedolizumab has been shown effective (e.g. 47% clinical response rate vs. 25% in placebo group) and is part of the current standard of care treatment in UC. With the observation of drastic increase of IBD patients in Asia, in which has historically low incidence of IBD, it is generally accepted that the westernized diet and urbanization of life style play an important role in IBD pathogenesis. Enteral nutritional therapy has been demonstrated effective in pediatric Crohn's disease (CD) patients; however, the application to adult IBD patients has not been widely accepted partly because of the compliance issue. In addition, unlike CD, neither enteral nutrition nor non-enteral nutrition in patients with active UC has been adequately studied. Therefore, this study proposes a novel approach to assess the integrated effect of a structured dietary intervention in active UC patients who will also be under the current standard of care medical therapy (vedolizumab). After this study achieves the proposed primary or secondary outcome, it will further support the hypothesized synergistic interactive therapeutic effect between the normalization of dysbiosis in the intestine (through dietary intervention) and anti-inflammatory biologics (vedolizumab).

DETAILED DESCRIPTION:
Specific Aims:

Hypothesis to be investigated: the integrated treatment effect of controlling inflammatory process through vedolizumab in active UC patients can be synergistically enhanced with a structured semi-vegetarian dietary intervention

Background and Significance:

Research of fecal microflora in UC has shown its influential role on the disease pathogenesis. In UC patients, the adaptive immune system is dysregulated and hyper-reactive to the commensal intestinal microﬂora in susceptible individuals and the diversity of intestinal ﬂora decreases, called dysbiosis, by 30% to 50%. For the treatment of moderate to severe UC, tumor necrosis factor (TNF) antagonists, although efficacious but predispose patients to serious infection. Vedolizumab, a humanized monoclonal antibody that specifically recognizes the α4β7 heterodimer, selectively blocking the migration of leukocytes into inflamed intestinal tissue, has been shown to achieve clinical response and clinical remission in patients with moderate to severely active UC (clinical response 47% vs. 25% (placebo) at week 6 and clinical remission 42% vs. 16% (placebo) at week 52) in patients with moderate to severely active UC. In epidemiological study, western diet characterized with high in animal fat and low in fruits and vegetables has been found associated with an increased risk of IBD. In murine models, diets high saturated animal fats has been shown to be associated with dysbiosis, increased intestinal permeability, decreased mucus layer, and increased release of pro-inflammatory cytokines. Additive in processed food, such as emulsifiers, has been recently found with impact on the mouse gut microbiota promoting colitis and metabolic syndrome. Enteral nutritional therapy has been demonstrated effective in pediatric IBD patients; however, the application to adult IBD patients has not been widely accepted partly because of compliance and adherence to the diet. Recently, non-enteral dietary interventions, such as semi-vegetarian diet, specific carbohydrate diet, and IBD exclusion diet, have gained attention based on small non-randomized trials. In a small prospective clinical trial in CD patients, semi-vegetarian diet was well tolerated and 93% (16 out of 17) of patients remained in clinical remission, compared with 33% (2 out of 6 patients) in an omnivorous diet group, at 2 years. A well-designed randomized clinical trial using a structured dietary intervention, which integrates the merits of previously proposed diets, is warranted, especially in conjunction with the current standard of care (e.g. vedolizumab) and the novel normalization of dysbiosis through structured semi-vegetarian dietary intervention.

Research Design and Methods:

Study Design or Overview:

This study is a pilot study of evaluating the synergistic effect of vedolizumab in conjunction with structured semi-vegetarian dietary intervention on the treatment of active UC patients who will be under the treatment of Vedolizumab. Subjects will be screened at outpatient clinic visit appointments and interested, qualified subjects will be consented and offered participation in this trial. Once consent has been obtained, baseline values will be established and subjects will begin treatment. A final visit for evaluation and collection of lab samples will be conducted at the end of the study at week 14.

Investigative Agent: vedolizumab in conjunction with semi-vegetarian dietary intervention:

Single interventional group: vedolizumab (300mg) IV infusions at week 0, 2, 6, 14 (as current standard of care) and concurrently on structured semi-vegetarian diet Duration of Therapy: 14 weeks; Duration of time on study: 14 weeks Structured semi-vegetarian dietary intervention (see supplementary material): Eligible study subjects will be counseled with a registered dietician and complete a Food Frequency Questionnaire to record and monitor the dietary pattern that the patient has at different time points, including prior to UC flare, current diet, diet during and after study.

The patient will be on a structured semi-vegetarian diet described below: (Specific recipes and food preparation will be provided during the counselling session with a dietician).

* Gradually increase calories, up to 25-30 kcals/kg/day
* Gradually add fiber (ex. white rice 2-5 days, then mixed rice 70% white to 30% brown rice) in an instructed regimen
* Daily vegetables, fruits, legumes, potatoes, probiotic food (miso, pickled vegetables), plain yogurt
* Encourage no smoking, regular physical exercise, moderate to no use of alcohol, regularity of meals, no snacking
* Foods to strictly limit/avoid: bread, cheese, margarine, fast foods, carbonated beverages, highly processed foods
* Diet excludes completely: Animal fat and Trans saturated fats, red meat and processed meat, sugar, emulsifiers (CMC, PS-80)

Sample Size:

Since this is a pilot study, no formal study power and sample size calculation is needed. The investigators plan to recruit 10 study subjects for the single interventional group.

Data Collection:

Clinical Assessments:

The primary outcome: Clinical response at week 6 (which is defined as ≥3 improvement in Mayo score (see page 4 for reference table), and a decrease of at least 30% from the baseline score).

The secondary outcome: Clinical response at week 14(which is defined as ≥3 improvement in Mayo score (see page 4 for reference table), and a decrease of at least 30% from the baseline score).

The investigators will also collect stool samples before (week -1) and after (week 14) the dietary interventions for microbiome study.

Data Analysis:

Univariate descriptive statistics and frequency distributions will be calculated, as appropriate for all variables including the primary and secondary outcomes. Baseline values for demographic, clinical, and outcome variables (primary and secondary) will be tabulated for the single interventional group. Primary outcome (clinical response rate at week 6) of this pilot study result will be non-analytically compared to the previously reported 47.1% from the previous clinical trial of vedolizumab alone in moderately to severe UC patients

Feasibility and Time Frame:

This is a pilot study and 10 study subjects will be enrolled by the end of 2017. Based on the current volume of eligible patients at the institution, it will be expected to complete the recruitment in 3 to 4 months. The completion of this study is estimated to be within 4 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* diagnosed with active UC (with a Mayo score ≥4, with an endoscopic Mayo Clinic score ≥1, and disease that extended 15 cm or more from the anal verge)
* failed with prior mesalamine therapy
* Patients who were previously exposed to mesalamine or steroids will have a 30-day washout period before being enrolled
* Patients who were previously exposed to tumor necrosis factor (TNF) antagonists will have a 60-day washout period before being enrolled
* For patients who were previously exposed to glucocorticoids, immunosuppressive medications (i.e., azathioprine, 6-mercaptopurine, or methotrexate), or TNF antagonists, a documentation of unsuccessful previous treatment (i.e., lack of response or unacceptable adverse events) is required
* A diagnosis of UC confirmed by biopsy obtained at the index colonoscopy or flexible sigmoidoscopy.

Exclusion Criteria:

* Patients who have been on semi-vegetarian diet before the trial will be excluded
* pregnancy or lactation
* an unstable or uncontrolled medical disorder
* an anticipated requirement for major surgery
* history of subtotal colectomy with ileorectostomy or colectomy with ileoanal pouch, Koch pouch, or ileostomy for UC, or planned bowel surgery
* unable to give informed consent
* current diagnosis of fulminant colitis or toxic megacolon, abdominal abscess, symptomatic colonic stricture, stoma
* disease limited to the rectum (ulcerative proctitis)
* current total parenteral nutrition
* positive Clostridium difficile stool assay
* history of an infection requiring intravenous antimicrobial therapy within 1 month or oral antimicrobial therapy within 2 weeks
* history of listeria, histoplasmosis, chronic or active hepatitis B or C infection, human immunodeficiency virus, immunodeficiency syndrome, untreated tuberculosis
* history of central nervous system demyelinating disease
* history of malignancy other than a successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix, or evidence of dysplasia or malignancy on the screening colonoscopy/flexible sigmoidoscopy with biopsy
* Any of the following laboratory abnormalities during the screening period:

  1. Hemoglobin level <8 g/dL
  2. WBC count <3 × 109/L
  3. Lymphocyte count <0.5 × 109/L
  4. Platelet count <100k/L or >1200k/L
  5. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 × the upper limit of normal (ULN)
  6. Alkaline phosphatase >3 × ULN, g) Serum creatinine >2 × ULN
* Antibiotic use within past 14 days; Probiotics use within past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical response at week 6 | 6 weeks
  Clinical response at week 6 (which is defined as ≥3 improvement in Mayo score, and a decrease of at least 30% from the baseline score).

SECONDARY OUTCOMES:
Clinical response at week 14 | 14 weeks
  Clinical response at week 14(which is defined as ≥3 improvement in Mayo score, and a decrease of at least 30% from the baseline score).

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Hsi Wang, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No